CLINICAL TRIAL: NCT04385706
Title: The Effectiveness of Joint Planning in Paediatric Rehabilitation: Parent and Child Related Outcomes
Brief Title: Joint Planning in Paediatric Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Western University, Canada (Other)
Responsible Party: Principal Investigator, Laura Brunton, Assistant Professor, Western University, Canada
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 115539
Record Dates: First submitted 2020-05-06; First posted 2020-05-13 (Actual); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Children With Developmental Delay

STUDY DESIGN:
Intervention Model Description: One group pre-test post-test design to evaluate a coaching model
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Applied Coaching Model (Experimental): One-group pre/post test
  Interventions: Behavioral: Applied Coaching Model

INTERVENTIONS:
Behavioral: Applied Coaching Model — The Applied Coaching Model incorporates key learning opportunities and coaching strategies with evidence-based practices, approaches and theories and will serve as a tool for all healthcare providers wanting to implement coaching techniques within their practice.

SUMMARY:
We will use one group, pretest-posttest research design. The intervention will have a 6-month timeframe. Up to 18 participants will be selected from active caseloads of the three to six participating healthcare providers in the Early Childhood Rehabilitation Program at the Alberta Children's Hospital, Child Development Centre site in Calgary Alberta. All data will be collected in Alberta using remote measures. Parents and therapists will complete surveys in an online portal. One measure needs to be completed in conjunction with the therapist and parent and will be done in person using an online portal. The researchers will have a local investigator (Debra Teitelbaum) in Calgary who works on-site to help manage data collection and recruitment in person if necessary.

ELIGIBILITY:
Inclusion Criteria:

* Receiving care for developmental delay

Exclusion Criteria:

* Cannot speak or read english

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 8 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Change in Canadian Occupational Performance Measure (COPM) | Change in COPM performance and satisfaction between baseline and 6-months.
  An evidence-based measure designed to capture a client's/familie's self-perception of performance in everyday living, their satisfaction with their performance, and changes in performance/satisfaction over time. It is one method of setting and measuring achievement of individualized therapeutic goals.

SECONDARY OUTCOMES:
Measure of Processes of Care (MPOC) | Change in MPOC (satisfaction) between baseline and 6-months.
  Satisfaction with healthcare services - the MPOC is a self-report measure of parents' perceptions of the extent to which the health services they and their child(ren) receive are family-centred.
PedsQL Family Impact Module | Change in PedsQL Family Impact Module between baseline and 6-months
  Quality of life
Parent Stress Index | Change in Parenting Stress Index between baseline and 6-months
  Stress
Self-efficacy Visual Analog Scale | Change in self-efficacy between baseline and 6-months
  self efficacy rating of ability to carry out home exercises, 0-100mm line, higher equals more self-efficacy
Therapist perceived parent efficacy Visual Analog Scale | Change in efficacy between baseline and 6-months
  Therapist rated parent efficacy rating of ability to carry out home exercises, 0-100mm line, higher equals more efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Laura K Brunton, PhD, Principal Investigator — Western University
Locations (1):
- Alberta Children's Hospital - Early Childhood Rehabilitation, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No
Individual participant data can be requested from the PI and all requests will be considered on an individual basis